CLINICAL TRIAL: NCT00601016
Title: A Phase II Study of Imiquimod 5 % Cream for the Treatment of Hemangioma in Infancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Graceway Pharmaceuticals, LLC (Industry)
Responsible Party: Catherine McCuaig, Pricipal Investigator, CHU Siante-Justine, CHU Sainte-Justine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-Mccuaig; 1
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Hemangioma, Capillary
Keywords: Infantile hemangioma; Hemangioma; Hemangioma of Infancy; benign tumors of infancy; Congenital hemangioma; Capillary
MeSH Terms: conditions — Hemangioma, Capillary; Hemangioma | interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Imiquimod 5% cream — Imiquimod 5% cream applied topical on hemangioma once a day , 3 to 7 times a week for a maximum of 4 months.
  Other Names: Imiquimod 5% cream = Aldara; Item ID = GH-6203-0328-5, CUP-051119552409; DIN number = 02239505; Lot number -= GFK026A

SUMMARY:
Hemangiomas of infancy, the most common benign tumors of infancy, are congenital or early infancy lesions characterized by a rapid postnatal growth, with high expression of angiogenic stimulators for 9-18 months, followed by slow regression for 5-9 years. Current therapies for the hemangiomas are usually restricted to more severe forms due to the risks of adverse effects, inconvenience and cost. Nevertheless, a substantial amount of the psychological discomfort and morbidity can be caused by untreated hemangiomas, especially those in the face.

Recently, Imiquimod 5% cream has emerged as a safe an effective drug for several skin conditions that benefit from modulation of the activity of the immune system, such as common warts and various forms of the skin pre-cancerous and cancerous lesions. Small case reports series have suggest that it could also be useful in hemangiomas, possibly through the inhibition of the angiogenesis by local IFN production.This is a small, open label study of 16 patients to document the efficacy of the Imiquimod 5% cream in the treatment of hemangioma of infancy (primary outcome). IFN and plasma drug levels, as well as clinical examinations and blood studies, will be carried out to evaluate safety of the treatment (secondary outcome). bFGF and VEGF will be measured in blood and urine in order to study the diagnostic and predictive value of these pro-angiogenic factors in the response of hemangiomas to the treatment with Imiquimod (secondary outcome).

The study is a phase II clinical trial of a once a day application of Imiquimod 5% cream, 3 to 7 times per week for a maximum of four months. The study held at the Dermatology Clinic of Sainte-Justine Hospital, and was completed within a 20 months timeframe after IRB approval.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants aged 2-12 months.
* Superficial or mixed hemangiomas in proliferative phase (growing in size in the last 1-2 months).
* Hemangiomas must be less than 10X10 cm and must not be ulcerated.

Exclusion Criteria:

* Preterm infant (less than 36 weeks of gestation).
* Ulceration of hemangioma prior to treatment.
* Immunosuppression.
* Hemangioma located on the eyelid or perianal region.
* Prior treatment of the hemangioma.
* Concomitant diseases.
* Presence of multiple hemangiomas and/or hemangiomas that would require systemic drug treatment.
* Potential difficulties with follow-up (patient from another town,difficult access to the hospital , etc.).
* History of allergy to any of the components of the drug preparation.
* Hemangiomas more than 10X 10 cm or ulcerated before the start of the treatment.

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2005-03; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To document the efficacy of Imiquimod 5% cream in the treatment of hemangioma of infancy. | Cream is applied for 4 months. Visits occured at month 1, 2, 4, and 8.

SECONDARY OUTCOMES:
IFN and plasma drug levels, as well as clinical examinations and blood studies, will be carried out to evaluate safety of the treatment. | 4 months of treatment. Doage done at each study visits (Month 1, 2 .4 and 8).
bFGF and VEGF will be measured in blood and urine in order to study the diagnostic and predictive value of these pro-angiogenic factors in the response of hemangiomas to the treatment with Imiquimod. | 4 months of treament with a follow-up at 8 months.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine McCuaig, M.D., Principal Investigator — St. Justine's Hospital
Locations (1):
- Sainte-Justine Hospital University Center (CHU), Montreal, Quebec, Canada

REFERENCES:
- [Background] Bruckner, A.L. and I.J. Frieden, Hemangiomas of infancy. J Am Acad Dermatol, 2003. 48(4): p. 477-93; quiz 494-6. 2. Dinehart, S.M., J. Kincannon, and R. Geronemus, Hemangiomas: evaluation and treatment. Dermatol Surg, 2001. 27(5): p. 475-85. 3. Jacobs, A.H. and R.G. Walton, The incidence of birthmarks in the neonate. Pediatrics, 1976. 58(2): p. 218-22. 4. Margileth, A.M. and M. Museles, Cutaneous hemangiomas in children. Diagnosis and conservative management. Jama, 1965. 194(5): p. 523-6. 5. Powell, T.G., et al., Epidemiology of strawberry haemangioma in low birthweight infants. Br J Dermatol, 1987. 116(5): p. 635-41. 6. Burton, B.K., et al., An increased incidence of haemangiomas in infants born following chorionic villus sampling (CVS). Prenat Diagn, 1995. 15(3): p. 209-14. 7. Martinez, M.I., et al., Infantile hemangioma: clinical resolution with 5% imiquimod cream. Arch Dermatol, 2002. 138(7): p. 881-4; discussion 884. 8. Gampper, T.J. and R.F. Morgan, Vascular anomalies: hemangiomas. Plast Reconstr Surg, 2002. 110(2): p. 572-85; quiz 586; discussion 587-8. 9. Ceisler, E.J., L. Santos, and F. Blei, Periocular hemangiomas: what every physician should know. Pediatr Dermatol, 2004. 21(1): p. 1-9. 10. Dadras, S.S., et al., Infantile hemangiomas are arrested in an early developmental vascular differentiation state. Mod Pathol, 2004. 17(9): p. 1068-79. 11. Oliver, G. and M. Detmar, The rediscovery of the lymphatic system: old and new insights into the development and biological function of the lymphatic vasculature. Genes Dev, 2002. 16(7): p. 773-83. 12. Vikkula, M., et al., Molecular basis of vascular anomalies. Trends Cardiovasc Med, 1998. 8(7): p. 281-92. 13. Cohen, M.M., Jr., Vasculogenesis, angiogenesis, hemangiomas, and vascular malformations. Am J Med Genet, 2002. 108(4): p. 265-74. 14. Chang, J., et al., Proliferative hemangiomas: analysis of cytokine gene expression and angiogenesis. Plast Reconstr Surg, 1999. 103(1): p. 1-9; discussion 10. 15. Takahashi, K., et al., Cellular markers that distinguish the phases of hemangioma during infancy and childhood. J Clin Invest, 1994. 93(6): p. 2357-64. 16. Bielenberg, D.R., et al., Progressive growth of infantile cutaneous hemangiomas is directly correlated with hyperplasia and angiogenesis of adjacent epidermis and inversely correlated with expression of the endogenous angiogenesis inhibitor, IFN-beta. Int J Oncol, 1999. 14(3): p. 401-8. 17. Ritter, M.R., et al., Insulin-like growth factor 2 and potential regulators of hemangioma growth and involution identified by large-scale expression analysis. Proc Natl Acad Sci U S A, 2002. 99(11): p. 7455-60. 18. Isik, F.F., et al., Monocyte chemoattractant protein-1 mRNA expression in hemangiomas and vascular malformations. J Surg Res, 1996. 61(1): p. 71-6. 19. Dosquet, C., et al., [Importance of bFGF (
- [Derived] McCuaig CC, Dubois J, Powell J, Belleville C, David M, Rousseau E, Gendron R, Jafarian F, Auger I. A phase II, open-label study of the efficacy and safety of imiquimod in the treatment of superficial and mixed infantile hemangioma. Pediatr Dermatol. 2009 Mar-Apr;26(2):203-12. doi: 10.1111/j.1525-1470.2008.00857.x. PMID 19419474